CLINICAL TRIAL: NCT05762562
Title: Parkinson Disease Telerehabilitation Program (PDTR): a Home-motor Program for Parkinson's Disease With Open-source Platforms. A Pilot Study.
Brief Title: Parkinson Disease Telerehabilitation Program (PDTR): a Home-motor Program. A Pilot Study.
Status: Completed | Type: Observational
Sponsor: Istituti Clinici Scientifici Maugeri SpA (Other)
Responsible Party: Principal Investigator, Chiara Vellata, Physiotherapy, Istituti Clinici Scientifici Maugeri SpA
Other Study IDs: prot. 2486 CE, 06/10/2020
Record Dates: First submitted 2023-01-11; First posted 2023-03-09 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Parkinson Disease
Keywords: Parkinson's Disease; Telerehabilitation; Remote Physical Activity; Rehabilitation; Digital Health
MeSH Terms: conditions — Parkinson Disease | interventions — Telerehabilitation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Telerehabilitation with OS platforms: Patients with Parkinson's Disease were divided into three subgruops based on their residual motor skills.
  Interventions: Other: Telerehabilitation with open source platforms

INTERVENTIONS:
Other: Telerehabilitation with open source platforms — Telerehabilitation with opensource platforms. Patients enrolled were dived into three groups based on their score in SPPB. Each group corresponded to a Program (Pr): • Pr. A is for patients with capable motor skills, Pr. B is for patients with reduced motor skills, • Pr. C is for patients who didn't show having sufficient motor skills to support a TR program. Patients who were included in TrP.A and TrP.B underwent a TR program using OS platforms for 8 consecutive weeks. A specific exercise program for the parkinsonian patients was structured in relation to the individual residual motor skills based on the FITT - frequency/intensity/type/time - protocol.
  Twice a week, the activity was performed with the support of a physiotherapist through OS TR platform.
  Subjects included in TmP.C participated in an 8-weeks program. A video-call was scheduled once a week to monitor the patient's clinical condition without any exercise program.

SUMMARY:
Parkinson's disease (PD) leads to multifactorial disabilities with consequent social restrictions, especially in the COVID-19 era. Continuity of care, especially rehabilitation measures, is critical to improve or maintain an adequate QoL for patients. The Parkinson Disease Telerehabilitation Program (PDTR) is an individualized home rehabilitation program using open-source platforms (OSp).

The main purpose of this pilot study is to investigate the feasibility of TR in patients with PD by using free OS platforms (PDTR PROGRAM).

The target of this study was to have at least 90% of participants completing the program. To complete the program every single patient had to complete at least 80% of the prescribed TR sessions.

DETAILED DESCRIPTION:
Participants were PD patient afferent to the Neurology ambulatory. Patients underwent an initial evaluation (T0) by the neurologist and physiotherapist. During T0, also the level of digital literacy was evaluated

Participants included in the study were separated into three groups based on their residual motor skills evaluated by the Short Physical Performance Battery (SPPB).

Each group corresponded to a Program (Pr). SPPB score between 12 and 10: Pr. A for patients with capable motor skills; they were were associated to the TR program A (TrP.A).

SPPB score between 9 and 7: Pr. B for patients with reduced motor skills; they were were associated to the TR program B (TrP.B).

SPPB score lower than 7: Pr. C for patients who didn't show having sufficient motor skills; they were were associated to the telemonitoring program C (TmP.C) without any exercise program.

Patients who were included in TrP.A and TrP.B underwent a TR program using OS platforms for 8 consecutive weeks.

OS platforms used are: Zoom, Skype, Google Teams, WhatsApp. The patient was given the opportunity to choose the operating system to use based on their knowledge, computer skills and ease of use to facilitate the management of the session.

Patients in TrP.A and TrP.B had to perform at home a tailored exercise program 4 times/week for 45-60 minutes.

Twice a week, the activity was performed with physiotherapist through OSp. A specific exercise program for the parkinsonian patients was structured in relation to the individual residual motor skills based on the FITT - frequency/intensity/type/time - protocol. Both programs, A and B, include multiple exercise: aerobic activities, mobility and stretching exercises for upper and lower limbs, global muscle strengthening, balance & motor coordination training, start and stop exercises and walking training.

The exercises in program A were more complex and showed a higher intensity, while those in program B were simpler, safer and at lower intensity.

Subjects included in TmP.C participated in an 8-weeks program. A video-call was scheduled once a week to monitor the patient's clinical condition without any exercise program.

The target of this study was to have at least 90% of participants completing the program. To complete the program every single patient had to complete at least 80% of the prescribed TR sessions.

ELIGIBILITY:
Inclusion Criteria:

* Hoehn & Yahr (H&Y) score between 1 and 3;
* being on drug treatment stabilized with L-Dopa or dopamine agonists;
* being able to walk independently (with or without help)
* having adequate computer knowledge, be able to use online communication platforms and to undertake a continuous 8-weeks program.

Exclusion Criteria:

* Montreal Cognitive Assessment screening test score below 17.54
* having unpredictable motor fluctuations or non-pharmacologically controlled dyskinesias
* having neurological pathologies superimposed on PD; or cognitive, sensory, psychiatric alterations such as to make it impossible to understand and execute the exercises; or musculoskeletal and cardiopulmonary diseases that compromise mild physical activity.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Parkinson's disease patients with different residual motor skills.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
The opportunity of the usage TR in PD patients by using free open-source platforms | 1 year
  90% of participants completing the program. To complete the program every single patient had to complete at least 80% of the prescribed TR sessions

SECONDARY OUTCOMES:
Patient's satisfaction | 1 year
  Administration of a specific questionnaire to evaluate the patient's satisfaction with TR treatment program with free open-source platforms
Patient's agreement | 1 year
  Administration of a specific questionnaire to evaluate the patient's agreement with TR treatment program with free open-source systems
Maintenance of clinical outcomes - Walking speed | 1 year
  Walking speed using 10 Meter Walking Test (10 MWT) rated in seconds. Comparison between T0 and T1 in the groups A and B. A descriptive analysis of the results was then conducted.
Maintenance of clinical outcomes - Balance | 1 year
  Balance using MiniBEST Test (values: 0 minimum - 28 maximum). Comparison between T0 and T1 in the groups A and B. A descriptive analysis of the results was then conducted.
Maintenance of clinical outcomes - Risk of falling | 1 year
  Risk of falling using the Time Up and Go (TUG Test) rated in seconds. Comparison between T0 and T1 in the groups A and B. A descriptive analysis of the results was then conducted.
Perceived level of quality of life | 1 years
  Evaluation of the level of perceived quality of life using the the Parkinson's Disease Questionnaire (short version)(PDQ-8), (values: 0 minimum - 32 maximum. The summed scor is then divided by total possible score an given as a percentage score out of 100). Comparison between T0 and T1 in the groups A and B.

CONTACTS AND LOCATIONS:
Locations (1):
- Ics Maugeri, Pavia, PV, Italy

IPD SHARING:
Plan to Share IPD: No